CLINICAL TRIAL: NCT06702059
Title: Cardiopulmonary Exercise Testing in the Prediction of Post-operative Complications in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Cardiopulmonary Exercise Testing in Cardiosurgery Patients
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Centre of Cardiovascular and Transplantation Surgery, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, Principal Investigator, St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: 46/2024/OD
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complications
Keywords: cardiovascular surgery; cardiopulmonary exercise testing; post-operative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- coronary artery bypass graft candidates: patients scheduled for CABG surgery will undergo pre-operative cardiopulmonary exercise testing and post-operative complications monitoring
  Interventions: Diagnostic Test: Cardiopulmonary exercise testing

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise testing — Subjects will undergo pre-operative cardiopulmonary exercise testing.

SUMMARY:
Cardiopulmonary exercise testing (CPET) is considered to be a gold standard in pre-operative risk assessment and stratification of high risk patients scheduled for major surgery. Surprisingly, only a limited number of studies examined the prognostic role of CPET in cardiothoracic surgery. This is in contrast with rather poor discriminating quality of cardiovascular surgery risk scores and predominantly elderly cardiovascular surgery patients, with significant comorbidity and high degree of frailty. Recently, CPET was shown feasible in coronary artery bypass grafting surgery candidates. Additionally, the rest parameter, which is the partial pressure of end-tidal carbon dioxide (PETCO2) and a submaximal exercise parameter (the VE/VCO2 slope) with good prognostic utility across multiple respiratory exchange ratio values), has been shown to predict mortality and post-operative complications.

Whether these rest and submaximal exercise parameters can be used to predict postoperative complications in cardiovascular surgery patients is yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for coronary artery bypass graft surgery

Exclusion Criteria:

* not able to perform cardiopulmonary exercise testing, off-pump revascularization, without full sternotomy, previous cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for coronary artery bypass graft surgery
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
post-operative pulmonary complications | within 30 post-operative days
  pneumonia, atelectasis, respiratory failure, ARDS
post-operative cardiovascular complications | within 30 post-operative days
  new arrhythmias (atrial fibrillation, supraventricular tachycardia, etc.), myocardial infarction/minimal myocardial lesion, hypotension, heart failure, pulmonary edema, pulmonary embolism, cardiopulmonary resuscitation

SECONDARY OUTCOMES:
Hospital and Intensive care length of stay | within 30 post-operative days
  Hospital and Intensive care length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, prof., M.D., Principal Investigator — St. Anne's University Hospital
Locations (2):
- Czechia (2):
  - Centre of Cardiovascular and Transplantation Surgery, Brno, Czech Republic
  - St. Anne's University Hospital in Brno, Brno, Czech Republic

IPD SHARING:
Plan to Share IPD: Undecided
Information will be provided upon reasonable request.

REFERENCES:
- [Background] Brat K, Tothova Z, Merta Z, Taskova A, Homolka P, Vasakova M, Skrickova J, Sramek V, Olson LJ, Cundrle I Jr. Resting End-Tidal Carbon Dioxide Predicts Respiratory Complications in Patients Undergoing Thoracic Surgical Procedures. Ann Thorac Surg. 2016 Nov;102(5):1725-1730. doi: 10.1016/j.athoracsur.2016.05.070. Epub 2016 Aug 3. PMID 27496629
- [Background] Cundrle I Jr, Merta Z, Bratova M, Homolka P, Mitas L, Sramek V, Svoboda M, Chovanec Z, Chobola M, Olson LJ, Brat K. The risk of post-operative pulmonary complications in lung resection candidates with normal forced expiratory volume in 1 s and diffusing capacity of the lung for carbon monoxide: a prospective multicentre study. ERJ Open Res. 2023 Mar 6;9(2):00421-2022. doi: 10.1183/23120541.00421-2022. eCollection 2023 Mar. PMID 36891072
- [Background] Mann J, Williams M, Wilson J, Yates D, Harrison A, Doherty P, Davies S. Exercise-induced myocardial dysfunction detected by cardiopulmonary exercise testing is associated with increased risk of mortality in major oncological colorectal surgery. Br J Anaesth. 2020 Apr;124(4):473-479. doi: 10.1016/j.bja.2019.12.043. Epub 2020 Feb 19. PMID 32085879
- [Background] Brunelli A, Belardinelli R, Pompili C, Xiume F, Refai M, Salati M, Sabbatini A. Minute ventilation-to-carbon dioxide output (VE/VCO2) slope is the strongest predictor of respiratory complications and death after pulmonary resection. Ann Thorac Surg. 2012 Jun;93(6):1802-6. doi: 10.1016/j.athoracsur.2012.03.022. Epub 2012 May 4. PMID 22560968
- [Background] Brat K, Homolka P, Merta Z, Chobola M, Heroutova M, Bratova M, Mitas L, Chovanec Z, Horvath T, Benej M, Ivicic J, Svoboda M, Sramek V, Olson LJ, Cundrle I Jr. Prediction of Postoperative Complications: Ventilatory Efficiency and Rest End-tidal Carbon Dioxide. Ann Thorac Surg. 2023 May;115(5):1305-1311. doi: 10.1016/j.athoracsur.2021.11.073. Epub 2022 Jan 21. PMID 35074321
- [Background] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266